CLINICAL TRIAL: NCT04930718
Title: Thumb and Wrist Proprioception Exercises to Improve Pain Sensibility and Manual Dexterity After Distal Radius Fracture.
Brief Title: Thumb and Wrist Proprioception Exercises.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Raquel Cantero-Téllez, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMA-Proprioception
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Radius Fractures; Hand Injuries; Pain, Chronic; Proprioceptive Disorders
MeSH Terms: conditions — Radius Fractures; Hand Injuries; Chronic Pain; Somatosensory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Wrist passive mobilizations; Actives exercises; Reeducation for Activity daily life;
  Interventions: Other: Thumb active Exercises
- Experimental group (Experimental): The experimental group will also carried out a proprioceptive exercise home program with a laptop.
  Interventions: Other: Thumb active Exercises

INTERVENTIONS:
Other: Thumb active Exercises — Active específico exercises; Reeducation program

SUMMARY:
Distal radius fracture is the most common upper extremity fracture with peak incidence among older women after the fifth decade of life. Proprioception is one constituent of a complex Sensory motor control process. Proprioception requires the reception and central integration of incoming afferent signals. Although various sensory and motor deficits have been correlated with significant functional impairment after wrist trauma, limited research exists on the effects of proprioception and multi sensory training after distal radius fracture.

DETAILED DESCRIPTION:
A randomized, controlled, single-center, double-blind, clinical trial, with 1:1 allocation ratio, will be carried out involving patients diagnosis of distal radius fracture (aged 18 years and above). Both assessor and statistician will remained blinded.

Standard rehabilitation program for distal radius fracture treatments will received for both the control and experimental groups for a period of 12 weeks. The experimental group, in addition, will received a proprioceptive training program during the same intervention period, which will be conducted twice weekly (24 sessions).

The severity of pain with activity will be measured according to the visual analog scale (VAS). PRWE questionnaire will be used to measure upper extremity function. Patient's occupational performance will be measured with the Canadian Occupational Performance Measure (COPM) and proprioception with Joint position sense (JPS) and force sense (FS) testing, for dexterity Due pegboard test will be used. All outcome measures will be collected at baseline, immediately following the intervention at 3 weeks and at 12 weeks following the end of the intervention.

Participation in the study will be voluntary and patients will be included if they satisfied specific inclusion criteria.

All procedures will be follow in accordance with the ethical standards of the responsible committee on human experimentation (institutional and national) and with the Helsinki Declaration. All participants will sign a written informed consent in accordance with guidelines approved by the local ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosis of distal radius fracture.
* Wrist immobilization after lesion (unless 3 weeks)
* Capacity for sing inform concept and understand the exercises

Exclusion Criteria:

* Others associate fractures in hand or upper limb
* Wrist ligaments injuries
* Neurological disorder affecting the upper limb
* Have received previous proprioceptive training for upper limb injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Joint position Sense (JPS) | baseline-3 months
  Proprioception using active joint position sense (JPS) has been utilized in studies to establish a correlation between therapy intervention and proprioception. Joint angle will be measured using a standard clear plastic goniometer.
Force sense (FS) | baseline-3 months
  Muscle strength (MS) is one of the most important factors affecting human performance. Force sense (FS) is also known as sense of effort / heaviness / tension or the force matching sense. It is the ability to reproduce (or match) a desired level of force one or more times.

SECONDARY OUTCOMES:
Pain (VAS) | baseline-3 months
  VAS has been shown to be a reliable and valid instrument for pain assessment which is used frequently for clinical and research purposes. It consists of a 10-cm line anchored at each end. The left-hand anchor reads 'no pain' and the right-hand anchor reads 'worst possible pain'; the patients marked a line to represent their pain level.
Canadian Occupational Performance Measure | baseline-3 months
  Patient's occupational performance will be measured with the Canadian Occupational Performance Measure (COPM). The COPM enables subjects to identify goals for hand therapy and engage in a subject-specific therapeutic process.
PRWE Patient review wrist evaluation | baseline-3 months
  PRWE is the Patient-Rated Wrist Evaluation, It is one of the reliable upper extremity outcome instrument.The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. Developed in 1998 for clinical assessment and is used for specific wrist problems.
Dexterity test. Purdue pegboard | baseline-3 months
  This manipulative dexterity test contains twenty-five holes with randomly positioned slots and pegs which have a key along one side. Pegs must be rotated to match the hole before they can be inserted.

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Cantero-Téllez, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided